CLINICAL TRIAL: NCT00068926
Title: VRC 300: Screening of Healthy Volunteers for Clinical Trials of Investigational Vaccines to Prevent Infectious Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030285; 03-I-0285
Record Dates: First submitted 2003-09-11; First posted 2003-09-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-29

CONDITIONS: Healthy
Keywords: Biodefense; Prevention; Emergent; Virus; Immune Response; Healthy Volunteer; HV
MeSH Terms: conditions — Virus Diseases

SUMMARY:
This protocol will screen healthy normal volunteers for participation in studies of vaccines under development at NIAID's Vaccine Research Center. Of interest are vaccines for:

* Newly identified infectious diseases such as SARS.
* Infectious diseases of concern as possible bioweapons, such as smallpox and Ebola virus
* Emerging infectious diseases that are more widespread geographically than in the past, such as West Nile virus
* For preventing diseases such as tuberculosis and malaria.

Healthy normal volunteers between 18 and 70 years of age may be eligible for this protocol. Screening begins about 1 to 6 months before the start of the vaccine study. Participants will have a physical examination and health history, including questions about sexual activity and drug use. Over the course of the screening visits, participants will be asked to give urine and blood samples to test for various infections and other medical problems. Women capable of getting pregnant will be given a pregnancy test. Women who are pregnant or breastfeeding will not be enrolled in the study.

At the end of the screening, participants will be informed about which vaccines are currently being tested in clinical trials for which they may be eligible. Once participants enroll in a vaccine study, their participation in the screening protocol ends.

DETAILED DESCRIPTION:
STUDY DESIGN: The purpose of the study is to screen potential study volunteers to determine if they are eligible for infectious disease vaccine clinical trials being sponsored by the Vaccine Research Center (VRC) at the NIH Clinical Center. All work will be conducted by the VRC Clinic of the National Institutes of Health or IRB-approved extramural sites that are collaborating with the VRC Clinic. Educational materials on vaccines will be reviewed with and provided to subjects before enrollment into the study.

SUBJECTS: Approximately 3,000 healthy adults; age 18-70 years.

STUDY DURATION: Duration of participation is variable, and may last from a few weeks to several months for each subject. Study participation is complete when the subject enrolls in a vaccine study, is found to be ineligible for all vaccine studies or declines to participate in any vaccine studies.

STUDY EVALUATIONS: Evaluations usually include history, physical examinations and laboratory tests. Only those evaluations needed to determine eligibility for a particular study will be done. Evaluations other than those described in this protocol may be done if necessary for eligibility for a study. Blood will also be collected for storage.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: 18 to 70 years of age

Available to participate for the planned duration of the investigational vaccine study for which the screening is being done (vaccine studies may require 6 months to 18 months of clinic visits).

Able and willing to complete the informed consent process.

Agree to have blood stored for future studies of the vaccine, the immune system, and/or other medical conditions.

EXCLUSION CRITERIA:

Known to be infected with HIV, syphilis, tuberculosis, hepatitis B or hepatitis C.

A condition in which repeated blood draws or injections pose more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access.

A condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being.

Known to be pregnant or breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 958 (Actual)
Dates: Start 2003-09-03; Study Completion 2011-06-29

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Clinical Alliance for Research and Education - Infectious Diseases, LLC, Annandale, Virginia

REFERENCES:
- [Background] Fauci AS. Infectious diseases: considerations for the 21st century. Clin Infect Dis. 2001 Mar 1;32(5):675-85. doi: 10.1086/319235. Epub 2001 Feb 23. PMID 11229834